CLINICAL TRIAL: NCT02893033
Title: Neuromodulation With rTMS in Dysphagic Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-07-007C
Record Dates: First submitted 2016-08-26; First posted 2016-09-08 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2016-07

CONDITIONS: Transcranial Magnetic Stimulation
Keywords: Dysphagia; Repetitive Transcranial Magnetic Stimulation; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real stimulation (Experimental): Real repetitive transcranial magnetic stimulation + swallowing training
  Interventions: Device: repetitive transcranial magnetic stimulation
- Sham stimulation (Sham Comparator): Sham repetitive transcranial magnetic stimulation + swallowing training
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — rTMS

SUMMARY:
The patients with chronic dysphagia secondary to first-ever stroke were randomly assigned to 2 groups: Group A: sham stimulation for 10 minutes , Group B: real rTMS for 10 minutes. rTMS conditioning: daily rTMS 10 min for 10 days. Assessments: 1. videofluoroscopy，2.Functional outcome swallowing scale (3 scales). 3. MEP measurements

DETAILED DESCRIPTION:
While the reﬂex component of swallowing depends on swallowing centres in the brainstem, initiation of swallowing is a voluntary action that involves the integrity of motor areas of the cerebral cortex. Oropharyngeal dysphagia occurs in more than 50% of stroke patients. Aspiration pneumonia occurs in up to 20% of acute stroke patients and is a major cause of mortality after discharge. Oropharyngeal dysphagia is both underestimated and underdiagnosed as a cause of major nutritional and respiratory complications in stroke patients. Recently, transcranial magnetic stimulation (TMS) has been used to study the cortical input to swallowing control and has revealed that the topographic representation of esophageal motor function in the human cerebral cortex is bilateral but with consistent interhemispheric asymmetry unrelated to handedness.

In a number of recent studies, poststroke motor and dysphagia performance has been improved after daily treatment sessions with repetitive TMS (rTMS) using an excitatory frequency in patients with hemispheric ischaemic stroke due to occlusion of territories of the middle cerebral artery. Our hypothesis was that rTMS would facilitate dysphagia recovery.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of stroke related dysphagia
2. no concurrent neurodegenerative or dementia history
3. an absence of TMS contraindications.

Exclusion Criteria:

* arrythmia, epilepsy, infection, hyperglycemia, pacemaker or implants, external ventricular drain or ventriculoperitoneal shunt

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
functional outcome | prior to treatment (baseline), on the next day after the 2 weeks treatment completion
  points of Australian Therapy Outcome Measures-the Swallowing scale as assessed by a clinical therapist

SECONDARY OUTCOMES:
videofluoroscopy | prior to treatment (baseline), on the next day after the 2 weeks treatment completion
  points of Penetration-Aspiration Scale as assessed by videofluoroscopy
cricopharyngeal motor evoked potentials | prior to treatment (baseline), on the next day after the 2 weeks treatment completion
  amplitude and latency measured by cricopharyngeal motor evoked potentials

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yi Tsai, Study Director — Department of Physical Medicine and Rehabilitation, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rofes L, Vilardell N, Clave P. Post-stroke dysphagia: progress at last. Neurogastroenterol Motil. 2013 Apr;25(4):278-82. doi: 10.1111/nmo.12112. Epub 2013 Mar 11. PMID 23480388
- [Background] Park JW, Oh JC, Lee JW, Yeo JS, Ryu KH. The effect of 5Hz high-frequency rTMS over contralesional pharyngeal motor cortex in post-stroke oropharyngeal dysphagia: a randomized controlled study. Neurogastroenterol Motil. 2013 Apr;25(4):324-e250. doi: 10.1111/nmo.12063. Epub 2012 Dec 23. PMID 23279198
- [Derived] Lin WS, Chou CL, Chang MH, Chung YM, Lin FG, Tsai PY. Vagus nerve magnetic modulation facilitates dysphagia recovery in patients with stroke involving the brainstem - A proof of concept study. Brain Stimul. 2018 Mar-Apr;11(2):264-270. doi: 10.1016/j.brs.2017.10.021. Epub 2017 Nov 7. PMID 29162502